CLINICAL TRIAL: NCT07077486
Title: A Randomized, Positvel Controlled, Multicenter Study of Effects of Telitacicept vs Cyclophosphamide on Lupus Realted Interstitial Lung Disease
Brief Title: Effects of Telitacicept vs Cyclophosphamide on Lupus Related Interstitial Lung Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Wuhan Central Hospital (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); Rongchang Biopharmaceutical (Unknown); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, YIKAI YU, the Deputy Chief Physician, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tongji Hospital
Record Dates: First submitted 2023-12-30; First posted 2025-07-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lupus or SLE; Interstitial Lung Disease; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lung Diseases, Interstitial | interventions — Methylprednisolone; Adrenal Cortex Hormones; Cyclophosphamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glucocorticoids and/or immunosuppressants other than CYC+ treatment with the Telitacicept group (Experimental): Telitacicept 160mg sc qw, plus standard of care therapy including glucocorticoids and/or immunosuppressants other than CYC sush as , tacrolimus, Sirolimus, cyclosporine, leflunomide, azathioprine, motecophenol ester, hydroxychloroquine, tripterine, methotrexate and sulazazopyridine. None of the cyclophosphamide usage was included in the group.
  Interventions: Drug: Methylprednisolone (Corticosteroid); Drug: Immunosuppressant other than CYC; Drug: Telitacicept Freeze-dried powder Injection 80mg
- glucocorticoids plus CYC and/or other immunosuppressants (Active Comparator): All patient in this group were administered with cyclophosphamide. The other immunosuppressants in this group include , tacrolimus, Sirolimus, cyclosporine, leflunomide, azathioprine, motecophenol ester, hydroxychloroquine, tripterine, methotrexate and sulazazopyridine. None of the biological agents like belimumab (Benlysta), anifrolumab (Saphnelo), telitacicept (TaiAi), tocilizumab (Actemra) and rituximab (Rituxan) was included in this group.
  Interventions: Drug: Methylprednisolone (Corticosteroid); Drug: Immunosuppressant other than CYC; Drug: Cyclophosphamide (CYC)

INTERVENTIONS:
Drug: Methylprednisolone (Corticosteroid) — In addition to conventional treatment (methyl-40mg or less /d), the treatment group also received hydroxychloroquine (100mg-200mg each time twice a day), and thalidomide (50mg-100mg each time once a day) could be added as appropriate.
  Other Names: Methyl
Drug: Immunosuppressant other than CYC — The control group only received conventional treatment (methyl 40 mg/d or less), and other traditional immunosuppressants (including but not limited to cyclophosphamide, tacrolimus, sirolimus, cyclosporine, leflunomide, azathioprine, motecophenol ester, hydroxychloroquine, tripterine, methotrexate and sulazazopyridine, etc.). No more than 3 types of immunosuppressant should be added during the whole treatment period, and the dose should not exceed 30% from the baseline period)
Drug: Telitacicept Freeze-dried powder Injection 80mg — Telitacicept is a TACI-Fc fusion protein, a type of drug used to treat autoimmune diseases. It works by targeting two key proteins, BLyS and APRIL, which are involved in the development and function of B cells, a type of white blood cell. By blocking these proteins, telitacicept can help to reduce B cell activity and suppress the immune system's overactivity in autoimmune diseases. Subcutaneous injection dose ranges from 80mg once a week to 160mg once a week.
  Arms: glucocorticoids and/or immunosuppressants other than CYC+ treatment with the Telitacicept group
Drug: Cyclophosphamide (CYC) — Cyclophosphamide iv injection is used for severe complications of systemic lupus erythematosus 400mg twice a week
  Arms: glucocorticoids plus CYC and/or other immunosuppressants

SUMMARY:
Recent data indicate that Telitacicept is beneficial for lupus nephritis. Our goal is to determine whether Telitacicept is an effective and safe treatment, compared to standard-of-care Cyclophosphamide, for subclinical and clinical ILD in patients with early lupus.

DETAILED DESCRIPTION:
Pulmonary abnormalities are present in up to 60% of patients with SLE, and up to 10% of the patients will develop clinical interstitial lung disease (ILD). Recent data indicate that Telitacicept is beneficial for lupus nephritis. Our goal is to determine whether Telitacicept is an effective and safe treatment, compared to standard-of-care Cyclophosphamide, for subclinical and clinical ILD in patients with early lupus. The study also explores disease mechanisms in lungs and serum immunological interaction, to identify potential biomarkers for diagnosis, prognosis, and response to treatment of lupus-ILD.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 2019 EULAR/ACR classification criteria for systemic lupus erythematosus;
* Male or non-pregnant female aged ≥ 18 years;
* Diagnosis by high-resolution lung CT (HRCT) is clearly consistent with interstitial lung disease (ILD);
* FEV1/FVC%≥60% and diffusion function DLCO (measured value/estimated value) ≥40%;
* Patients voluntarily participate in this trial, have good compliance, and have the ability to understand and sign informed consent before the study.

Exclusion Criteria:

* Alanine aminotransferase and/or aspartate aminotransferase (ALT/AST) > 5 times the upper limit of normal;
* severe chronic kidney disease (stage IV) or need for dialysis (estimated glomerular filtration rate (eGFR) < 30ml/min/1.73m2);
* Hemoglobin < 80 g/L;
* WBC < 2.0×10^9;
* Platelet < 50×10^9;
* Is pregnant or breastfeeding;
* Expected transfer to another hospital in a non-study site within 4 weeks (possibility of loss to follow-up);
* Life expectancy does not exceed 24 weeks;
* Have a history of severe allergies;
* Patients with other serious lung diseases or other clinically significant serious abnormalities in the lungs;
* Are using antitumor drugs, other immunosuppressants or immunomodulatory therapies;
* Significant pulmonary hypertension;
* Previous clinical or echocardiographic evidence of significant right heart failure;

  1. Right heart catheterization showing cardiac index ≤ 2 L/min/m2;
  2. Pulmonary hypertension requiring treatment with epoprostenol/traprostacyclin.
* Patients with severe cardiovascular disease:

  1. myocardial infarction within 6 months;
  2. Unstable angina within 6 months.
* Risk of bleeding, any of the criteria listed below:

  1. known genetic predisposition to bleeding;
  2. Patients who require the following treatments:

  i. Fibrinolytic therapy, full-dose therapeutic anticoagulation (e.g., vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin); ii. High-dose antiplatelet therapy. [Note: Prophylactic low-dose heparin or heparin flush solution (e.g., enoxaparin, 4000 I.U. S.C. per day) required for maintenance of indwelling intravenous access devices is not prohibited.) and prophylactic antiplatelet therapy (e.g., acetylsalicylic acid up to 325 mg/day, or clopidogrel at a dose of 75 mg/day, or other antiplatelet therapy at the same dose).
* History of hemorrhagic central nervous system (CNS) events within 12 months;
* Any of the following conditions within a period of 3 months:

  1. hemoptysis or hematuria;
  2. Active gastrointestinal bleeding or gastrointestinal ulcers;
* Have previously undergone hematopoietic stem cell transplantation (HSCT), or plan to receive HSCT in the following year, or plan to undergo major surgery.
* Women who are pregnant, breastfeeding or planning to become pregnant during the test;
* 28 days before administration or 3 months after administration, women of childbearing age are unwilling or unable to use highly effective contraceptive methods;
* According to the investigator's point of view, the patient has alcohol or drug abuse;
* History of dysphagia or any gastrointestinal disease that affects drug
* Patients with contraindications to the use of tatacept;
* Subjects deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Correlation between change from baseline at week 52 in forced vital capacity (FVC) [percentage (%) predicted] | At baseline and at week 24, 52
  Pulmonary function measurement (FEV1/FVC% % post-treatment difference during baseline)

SECONDARY OUTCOMES:
Correlation between change from baseline at week 52 in diffusing capacity for carbon monoxide (DLco) [percentage (%) predicted] | At baseline and at week 24, 52
  Diffuse function DLco measurement (% post-treatment difference at baseline)
Anti-double-stranded DNA antibody conversion ratio | At baseline and at week 12, 24, and 52
  Anti-double-stranded DNA antibody conversion ratio
Complement C3 and C4 levels return to normal ratios | At baseline and at week 12, 24, and 52
  Complement C3 and C4 levels return to normal ratios
Six minutes walking distance | At baseline and at week 12, 24, and 52
  The 6-minute walk test (6MWT) is a simple, submaximal exercise test commonly used to assess functional capacity in individuals with interstitial lung disease (ILD). It measures the distance a person can walk in six minutes, and this distance (6MWD) can be correlated with disease severity and prognosis.
Changes from baseline in cumulative corticosteroid dose at week 52 | At baseline and at week 52
  Baseline dose was defined as the average corticosteroid dose (prednisone equivalent for all oral, IV, subcutaneous [SC], or intramuscular [IM] administrations) over the 7 days prior to, but not including, day 0; this was used to model the normalized cumulative baseline dose over 52 weeks. Actual cumulative corticosteroid dose (prednisone equivalent for all oral, IV, SC, or IM administrations) over 52 weeks was calculated
Krebs von den Lungen-6 | At baseline and at week 12, 24, and 52
  Krebs von den Lungen-6 (KL-6), is a biomarker primarily associated with interstitial lung disease (ILD). It's a high-molecular-weight mucin-like glycoprotein produced by type II alveolar pneumocytes. Elevated KL-6 levels in the blood can indicate the presence, severity, and progression of ILD.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China